CLINICAL TRIAL: NCT04807153
Title: Exercise Capacity, Pulmonary Function and Physical Activity Levels in Patients With Lung Cancer Undergoing Pneumonectomy
Brief Title: Exercise Capacity, Pulmonary Function and Physical Activity Level in Patients Lung Cancer Undergoing Pneumonectomy
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Prof. Dr., Gazi University
Other Study IDs: Gazi University 23
Record Dates: First submitted 2021-02-28; First posted 2021-03-19 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Pneumonectomy; Status
Keywords: Lung Cancer; Pneumonectomy; Exercise Capacity; Upper Extremity Exercise Capacity; Physical Activity; Pulmonary Function
MeSH Terms: conditions — Lung Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Functional exercise capacity (6 minutes walk test), upper extremity exercise capacity (6 minutes Pegboard and Ring Test), respiratory functions (spirometer), respiratory muscle strength (mouth pressure measurement), peripheral muscle strength (dynamometer), respiratory muscle endurance (incremental threshold loading test), physical activity level (multi-sensor activity monitor), quality of life (European Cancer Research and Treatment Organization Quality of Life Scale (EORTC QOL C-30)), fatigue (Fatigue Severity Scale) and shortness of breath (Modified Medical Research Council (MMRC)) will be evaluated.
- Healthy Controls: Functional exercise capacity (6 minutes walk test), upper extremity exercise capacity (6 minutes Pegboard and Ring Test), respiratory functions (spirometer), respiratory muscle strength (mouth pressure measurement), peripheral muscle strength (dynamometer), respiratory muscle endurance (incremental threshold loading test), physical activity level (multi-sensor activity monitor), quality of life (European Cancer Research and Treatment Organization Quality of Life Scale (EORTC QOL C-30)), fatigue (Fatigue Severity Scale) and shortness of breath (Modified Medical Research Council (MMRC)) will be evaluated.

SUMMARY:
Pneumonectomy is a high-risk surgical procedure, causing impaired respiratory functions and exercise intolerance. It is associated with decreased physical activity, quality of life and increased fatigue.

The primary aim of the study is to compare the exercise capacity and respiratory functions of lung cancer patients undergoing pneumonectomy and healthy individuals. The secondary aim of the study is to compare peripheral and respiratory muscle strength, respiratory muscle endurance, physical activity level, shortness of breath, fatigue and quality of life of lung cancer patients undergoing pneumonectomy and healthy individuals.

DETAILED DESCRIPTION:
Pneumonectomy is a high risk surgical procedure compared to lobectomy, segmentectomy and non-anatomical resection. Pneumonectomy causes impairment of respiratory functions and exercise intolerance. Assessment of exercise capacity in pneumonectomy is prognostically important. Exercise intolerance can also occur with daily activities using the upper extremity. There is no study investigated upper extremity exercise capacity in this patient population. Postoperative pulmonary functions are determinant for early postoperative results as well as long-term postoperative quality of life. Therefore, it is necessary to evaluate respiratory functions in patients after surgery. Respiratory muscle functions are impaired due to changes in chest wall mechanics and incisions applied to respiratory muscles after surgery. There is no study investigated respiratory muscle endurance in this patient population.

Pneumonectomy is associated with decreased physical activity and quality of life. The number of studies investigating physical activity level in lung cancer patients undergoing pneumonectomy is limited. In this study, physical activity level will be evaluated by metabolic holter. Pneumonectomy has been shown as a predictor of deterioration in quality of life after surgery. In this study, the quality of life will be evaluated using a questionnaire specific to the disease. Fatigue is a common symptom in patients after lung cancer surgery. It negatively affects the patients quality of life and long-term prognosis.

Lung cancer patients undergoing pneumonectomy by the physicians of Gazi University Thoracic Surgery Department and healthy individuals will be included in this study. Patients and healthy individuals will be evaluated and the evaluation results will be compared. According to the sample size analysis 17 patients and 17 healthy individuals with similar demographic characteristics will be included the study. Patients and healthy individuals will be selected according to predetermined inclusion and exclusion criteria. The assessments will be completed in two days.

Functional exercise capacity (6 minutes walk test), upper extremity exercise capacity (6 minutes Pegboard and Ring Test), respiratory functions (spirometer), respiratory muscle strength (mouth pressure measurement), peripheral muscle strength (dynamometer), respiratory muscle endurance (incremental threshold loading test), physical activity level (multi-sensor activity monitor), quality of life (European Cancer Research and Treatment Organization Quality of Life Scale (EORTC QOL C-30)), fatigue (Fatigue Severity Scale) and shortness of breath (Modified Medical Research Council (MMRC)) will be evaluated.

ELIGIBILITY:
Inclusion criteria for patients group: Patients who are;

* pneumonectomy for lung cancer
* at least 6 weeks and at most 5 years after surgery
* being between ages of 20 and 80
* one of video-assisted thoracoscopic surgery or open thoracic surgery

Exclusion criteria for patients group: Patients who are;

* having comorbidities such as uncontrolled hypertension, diabetes mellitus, heart failure or atrial fibrillation
* having health problems such as cooperation
* having acute infection during evaluation
* having orthopedic, neurological, psychological, etc. problems that limit evaluations

Inclusion criteria for healthy group: Participants who are;

* willing to participate to the study
* being between ages of 20 and 80

Exclusion criteria for healthy group: Participants who are;

* having any diagnosis of chronic diseases
* having health problems such as cooperation
* having acute infection during evaluation
* being current smokers
* being ex-smokers (≥10 pack*years)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At least 17 patients with lung cancer patients undergoing pneumonectomy will be included in patients group and 17 healthy individuals will be included in control group
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Functional Exercise Capacity | First Day
  Functional exercise capacity will be evaluated with 6-minute walking test according to the American Thoracic Society and European Respiratory Society criteria.
Upper Extremity Exercise Capacity | First Day
  The functional capacity of the upper extremities will be evaluated with a six-minute pegboard and ring test (6-PBRT). Subjects are asked to move as many rings as possible in 6 minutes. The score is the number of rings moved during the 6-minute period.
Pulmonary function (Forced vital capacity (FVC)) | First Day
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, forced vital capacity (FVC) will be evaluated.
Pulmonary function (Forced expiratory volume in the first second (FEV1)) | First Day
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, forced expiratory volume in the first second (FEV1) will be evaluated.
Pulmonary function (FEV1 / FVC) | First Day
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, FEV1 / FVC will be evaluated.
Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) | First Day
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, flow rate 25-75% of forced expiratory volume (FEF 25-75%) will be evaluated.
Pulmonary function (Peak flow rate (PEF)) | First Day
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, peak flow rate (PEF) will be evaluated.

SECONDARY OUTCOMES:
Respiratory Muscle Strength | First Day
  Maximal inspiratory and expiratory muscle strength will be evaluated using mouth pressure device.
Peripheral Muscle Strength | Second Day
  Shoulder abduction and knee extensor muscle strength using portable hand held dynamometer will be evaluated.
Respiratory Muscle Endurance | First Day
  Respiratory muscle endurance will be assessed by the POWERbreathe Wellness (POWERbreathe, Inspiratory Muscle Training (IMT) Technologies Ltd., Birmingham, UK) device and the respiratory muscle endurance test at increased threshold load.
  The test will be started with 30% of the maximal inspiratory pressure and the pressure will be increased to 40%, 50%, 60%, %70, 80% 90% and 100% every two minutes. Patients will be asked to continue breathing through the device during the test. During the test, the number of breaths delivered during each 2-minute period will be recorded. If the individual cannot breathe 3 consecutive times, the test will be terminated by the physiotherapist.
  The total duration of the test and the maximum pressure value at which it continues to breathe for at least 1 minute will be multiplied. The value found will be recorded as the respiratory muscle endurance value.
Physical Activity Level | Second Day
  Physical activity will be evaluated using multi sensor activity monitor.
Disease Specific Quality of Life | Second Day
  Quality of life will be measured using Turkish version of European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 version 3.0 (EORTCQLQ).
  The cancer-specific questionnaire has 30 questions and incorporates five functional scales, three symptom scales, a global health status and several single items. All item scores are transformed to 0-100. Higher values indicate higher functional/health level in functional scales, a higher quality of life level in global health status and increased symptoms in symptom scales.
Fatigue | Second Day
  Fatigue will be evaluated using Turkish version of Fatigue Severity Scale. This questionnaire includes 9 items and score range for each item from 1 to 7 point (7-point Likert scale). Fatigue Severity Scale score is calculates by deriving an arithmetic mean. Cut-scores of over 4 are indicative of significant fatigue (higher scores show more severe fatigue).
Shortness of breath | First Day
  The Modified Medical Research Council (MMRC) dyspnea scale will be used to determine the perception of dyspnea during activities of daily living.
  Dyspnea is graded as: zero (shortness of breath with strenuous exercise only); one (shortness of breath when rushing or walking up a slight uphill); two (because of shortness of breath they walk slower than people of the same age or have to stop to breathe while walking at their own pace); three (stops to breathe after walking 100 meters or after a few minutes); and four (too short of breath to leave the house or shortness of breath when getting dressed).

CONTACTS AND LOCATIONS:
Overall Officials: Meral BOŞNAK GÜÇLÜ, Prof.Dr., Study Director — Gazi University; Gülsüm SERTTAŞ, Study Chair — Gazi University; Nur Dilvin ÖZKAN, MD, Principal Investigator — Gazi University; Ali ÇELİK, Assoc. Prof., Principal Investigator — Gazi University; İsmail Cüneyt KURUL, Prof.Dr., Principal Investigator — Gazi University
Locations (1):
- Gazi University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Unit, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vainshelboim B, Fox BD, Saute M, Sagie A, Yehoshua L, Fuks L, Schneer S, Kramer MR. Limitations in exercise and functional capacity in long-term postpneumonectomy patients. J Cardiopulm Rehabil Prev. 2015 Jan-Feb;35(1):56-64. doi: 10.1097/HCR.0000000000000085. PMID 25350720
- [Background] Deslauriers J, Ugalde P, Miro S, Deslauriers DR, Ferland S, Bergeron S, Lacasse Y, Provencher S. Long-term physiological consequences of pneumonectomy. Semin Thorac Cardiovasc Surg. 2011 Autumn;23(3):196-202. doi: 10.1053/j.semtcvs.2011.10.008. PMID 22172356
- [Background] Brocki BC, Westerdahl E, Langer D, Souza DSR, Andreasen JJ. Decrease in pulmonary function and oxygenation after lung resection. ERJ Open Res. 2018 Jan 19;4(1):00055-2017. doi: 10.1183/23120541.00055-2017. eCollection 2018 Jan. PMID 29362707
- [Background] Menna C, Ciccone AM, Ibrahim M, Andreetti C, D'Andrilli A, Maurizi G, Cassiano F, Cavaliere I, Venuta F, Rendina EA. Pneumonectomy: quality of life and long-term results. Minerva Chir. 2012 Jun;67(3):219-26. English, Italian. PMID 22691825
- [Background] Agostini PJ, Naidu B, Rajesh P, Steyn R, Bishay E, Kalkat M, Singh S. Potentially modifiable factors contribute to limitation in physical activity following thoracotomy and lung resection: a prospective observational study. J Cardiothorac Surg. 2014 Sep 27;9:128. doi: 10.1186/1749-8090-9-128. PMID 25262229
- [Derived] Serttas Guven G, Ozkan Koyuncuoglu ND, Celik A, Kurul IC, Bosnak Guclu M. Upper extremity functional exercise capacity, muscle oxygenation, respiratory muscle strength, and physical activity levels in patients underwent pneumonectomy for lung cancer: a cross-sectional study. Support Care Cancer. 2025 Aug 1;33(8):739. doi: 10.1007/s00520-025-09731-z. PMID 40748386